CLINICAL TRIAL: NCT01557257
Title: An Open-label, Single-dose and Multiple-dose, Randomized, Crossover Study to Evaluate Pharmacokinetics, Safety and Tolerability After Administration of ALO-02 40 Mg Twice Daily Compared to ALO-02 80 Mg Once Daily and to Oxycontin 40 Mg Twice Daily in Healthy Volunteers
Brief Title: Pharmacokinetics Study of ALO-02 and OxyContin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B4531006
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Management of Moderate to Severe Pain
Keywords: single- and multiple-dose pharmacokinetics; ALO-02; OxyContin
MeSH Terms: interventions — oxycodone naltrexone combination; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 40 mg ALO-02 capsule (Experimental): Single- and multiple-dose of 40 mg ALO-02 capsule under 50 mg naltrexone block
  Interventions: Drug: ALO-02; Drug: Naltrexone block
- 80 mg ALO-02 capsule (Experimental): Single- and multiple-dose of 80 mg ALO-02 capsule under 50 mg naltrexone block
  Interventions: Drug: ALO-02; Drug: Naltrexone block
- 40 mg OxyContin tablet (Experimental): Single- and multiple-dose of 40 mg OxyContin tablet under 50 mg naltrexone block
  Interventions: Drug: OxyContin; Drug: Naltrexone block

INTERVENTIONS:
Drug: ALO-02 — Day 1 (40 mg ALO-02 capsule, single dose) Days 2-5 (40 mg ALO-02 capsule, twice daily)
  Arms: 40 mg ALO-02 capsule
Drug: Naltrexone block — Naltrexone Hcl 50 mg tablet will be administered (1) 12.5 hours prior to, 30 minutes prior to, and 11.5 hours after Day 1 dosing, (2) 30 minutes prior to each dose of study drug on Days 2-5 dosing, (3) 11.5 hours after Day 5 PM dosing
  Arms: 40 mg ALO-02 capsule
Drug: ALO-02 — Day 1 (80 mg ALO-02 capsule, single dose) Days 2-5 (80 mg ALO-02 capsule, once daily)
  Arms: 80 mg ALO-02 capsule
Drug: Naltrexone block — Naltrexone Hcl 50 mg tablet will be administered (1) 12.5 hours prior to, 30 minutes prior to, and 11.5 hours after Day 1 dosing, (2) 30 minutes prior to each dose and 11.5 hours after the AM dosing on Days 2-5, (3) 23.5 hours after Day 5 dosing.
  Arms: 80 mg ALO-02 capsule
Drug: OxyContin — Day 1 (40 mg OxyContin tablet, single dose) Days 2-5 (40 mg OxyContin tablet, twice daily)
  Arms: 40 mg OxyContin tablet
Drug: Naltrexone block — Naltrexone Hcl 50 mg tablet will be administered (1) 12.5 hours prior to, 30 minutes prior to, and 11.5 hours after Day 1 dosing, (2) 30 minutes prior to each dose of study drug on Days 2-5 dosing, (3) 11.5 hours after Day 5 PM dosing
  Arms: 40 mg OxyContin tablet

SUMMARY:
To characterize the single- and multiple-dose pharmacokinetics of oxycodone following the administration of ALO-02 40 Mg Twice Daily, ALO-02 80 Mg Once Daily or Oxycontin 40 Mg Twice Daily in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive.

Exclusion Criteria:

* Evidence or history of clinically significant diseases.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Single-dose administration: Maximum Observed Plasma Concentration (Cmax) of oxycodone | 0, 1, 2, 4, 6, 8, 12, 14, 16, and 24 hours post Day 1 dosing
Single-dose administration: Area under the plasma concentration versus time curve from time zero to 24 hours (AUC24) of oxycodone | 0, 1, 2, 4, 6, 8, 12, 14, 16, and 24 hours post Day 1 dosing
Single-dose administration: Time to Reach Maximum Observed Plasma Concentration (Tmax) of oxycodone | 0, 1, 2, 4, 6, 8, 12, 14, 16, and 24 hours post Day 1 dosing
Multiple-dose administration: Area under the plasma concentration versus time curve from time zero to 24 hours (AUC24) of oxycodone, as data permit. | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing
Multiple-dose administration: Area under the plasma concentration versus time curve within a dosing interval of τ at steady state (AUCτ) of oxycodone, as data permit. | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing
Multiple-dose administration: Maximum plasma concentration at steady state on Day 5 (Cmax,ss) of oxycodone, as data permit. | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing
Multiple-dose administration: Minimum plasma concentration at steady state on Day 5 (Cmin,ss) of oxycodone, as data permit. | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing
Multiple-dose administration: Average plasma concentration at steady state on Day 5 (Cave,ss) of oxycodone, as data permit. | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing
Multiple-dose administration: Time to Reach Maximum Observed Plasma Concentration on Day 5 (Tmax) of oxycodone, as data permit. | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing
Multiple-dose administration: Plasma Decay Half-Life (t1/2) of oxycodone, as data permit. | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing
Multiple-dose administration: Peak to trough fluctuation at steady state (PTF) of oxycodone, as data permit. | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing
Multiple-dose administration: Accumulation ratio based on Area Under Curve (AUC) (Rac) of oxycodone, as data permit. | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing

SECONDARY OUTCOMES:
Single-dose administration: Dose normalized Maximum Observed Plasma Concentration (Cmax(dn)) of oxycodone, noroxycodone, and oxymorphone. | 0, 1, 2, 4, 6, 8, 12, 14, 16, and 24 hours post Day 1 dosing
Single-dose administration: Dose-normalized Area under the plasma concentration versus time curve from time zero to 24 hours (AUC24(dn)) of oxycodone, noroxycodone, and oxymorphone. | 0, 1, 2, 4, 6, 8, 12, 14, 16, and 24 hours post Day 1 dosing
Single-dose administration: Maximum Observed Plasma Concentration (Cmax) of noroxycodone and oxymorphone. | 0, 1, 2, 4, 6, 8, 12, 14, 16, and 24 hours post Day 1 dosing
Single-dose administration: Area under the plasma concentration versus time curve from time zero to 24 hours (AUC24) of noroxycodone and oxymorphone. | 0, 1, 2, 4, 6, 8, 12, 14, 16, and 24 hours post Day 1 dosing
Single-dose administration: Time to Reach Maximum Observed Plasma Concentration (Tmax) of noroxycodone and oxymorphone. | 0, 1, 2, 4, 6, 8, 12, 14, 16, and 24 hours post Day 1 dosing
Multiple-dose administration: Accumulation ratio (Rac) of oxycodone, as data permit | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing
Multiple-dose administration: Maximum Observed Plasma Concentration (Cmax) of oxycodone, as data permit | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing
Multiple-dose administration: Area under the plasma concentration versus time curve from time zero to 24 hours (AUC24) of noroxycodone and oxymorphone, as data permit. | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing
Multiple-dose administration: Area under the plasma concentration versus time curve within a dosing interval of τ (AUCτ) of noroxycodone and oxymorphone, as data permit. | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing
Multiple-dose administration: Maximum plasma concentration at steady state (Cmax,ss) of noroxycodone and oxymorphone, as data permit. | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing
Multiple-dose administration: Minimum plasma concentration at steady state (Cmin,ss) of noroxycodone and oxymorphone, as data permit. | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing
Multiple-dose administration: Average plasma concentration at steady state (Cave,ss) of noroxycodone and oxymorphone, as data permit. | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing
Multiple-dose administration: Time to Reach Maximum Observed Plasma Concentration (Tmax) of noroxycodone and oxymorphone, as data permit. | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing
Multiple-dose administration: Plasma Decay Half-Life (t1/2) of noroxycodone and oxymorphone, as data permit. | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing
Multiple-dose administration: Peak to trough fluctuation at steady state (PTF) of noroxycodone and oxymorphone, as data permit. | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing
Multiple-dose administration: Rac of noroxycodone and oxymorphone, as data permit. | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing
Multiple-dose administration: Maximum Observed Plasma Concentration (Cmax) of noroxycodone and oxymorphone, as data permit. | 96,96.5,97,98,100,102,104,108,108.5,109,110,112,114,116,120,132,144,168 hours post Day 1 dosing

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4531006&StudyName=Pharmacokinetics%20Study%20of%20ALO-02%20and%20OxyContin%0A